CLINICAL TRIAL: NCT01310608
Title: Effect of Preoperative Imaging of the Ascending Aorta With Modified Transoesophageal Echocardiography on New Dw-MRI Lesions After Cardiac Surgery
Brief Title: Effect Study of Modified Transoesophageal Echocardiography on Cerebral Embolization After Cardiothoracic Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Isala (Other)
Collaborators: Zorgvernieuwing (Other)
Responsible Party: Principal Investigator, Arno P. Nierich, MD. PhD, Isala
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: A-View 3
Record Dates: First submitted 2011-03-07; First posted 2011-03-08 (Estimated); Last update posted 2012-08-09 (Estimated); Status verified 2012-08

CONDITIONS: Coronary Artery Atherosclerosis
Keywords: Atherosclerosis aorta; A-View; Distal ascending aorta; Transoesophageal echocardiography; CABG; Cerebral embolisation
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A-View (Experimental)
  Interventions: Other: A-View
- No A-View (No Intervention)

INTERVENTIONS:
Other: A-View — Pre-operative imaging of the thoracic aorta with A-View technique
  Other Names: The A-View®; Aortic-view®; Modified transoesophageal echocardiography; FDA: 070515
  Arms: A-View

SUMMARY:
Patients undergoing cardiac surgery frequently develop neurologic complications, ranging from subtle cognitive changes to evident confusion, delirium, and stroke. This continuum of complications is commonly caused by embolization in the brain due to manipulation of atherosclerotic parts of the aorta ascendens (AA) during surgery. Timely detection of AA atherosclerosis before surgery enables the surgeon to consider changes of the surgical plan, to reduce the risk of embolization and thus subsequent neurologic complications.

Various methods exist to visualize the AA to detect atherosclerosis. Epiaortic ultrasound scanning has become the gold standard, but is seldom used as it interferes often with surgical plan and can only be used after sternotomy. Transesophageal echocardiography (TEE) is a widely used imaging method permitting evaluation of the aorta preoperatively, but assessment of distal AA is hampered by interposition of air-filled trachea between esophagus and AA. The A-View® (Aortic-view) method, a modification of conventional TEE using a fluidfilled balloon, overcomes this limitation. The safety and diagnostic accuracy of the A-View® have successfully been shown in previous studies. The hypothesis of this study is that the use of A-View will reduce cerebral embolization secondary to a change of surgical technique.

ELIGIBILITY:
Inclusion Criteria:

* Isolated CABG
* Elective surgery
* Stroke Risk Index <75(Newman, '96)

Exclusion Criteria:

* Other than isolated CABG
* Contra-indication for TEE
* Contra-indication for A-View
* Contra-indication for MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2011-03; Primary Completion 2011-03 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
New diffusion-weighted lesions on cerebral MRI | 3 - 4 Days after intervention

SECONDARY OUTCOMES:
The number, size, and location of new ischemic lesions on the postoperative DW-MRI | 3 - 4 Days after intervention
Any neurologic event during the first six postoperative weeks, which is manifested as either stroke, or transient ischemic attack (TIA), epileptic insults, or delirium, or cognitive deficit | 6 weeks postoperative
Stroke or TIA during the first three postoperative months | 3 months postoperative
Delirium during hospital stay | Until hospital discharge
Quality of life | 6 weeks and 1 year after the intervention
Number of "HITS" detected by Transcranial Doppler | peroperive
Incidence of Near Infrared Spectrography desaturations (NIRO 2000) | Peroperative
Short psychometric test | 6 weeks after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Arno Nierich, MD, PhD, Principal Investigator — Isala